CLINICAL TRIAL: NCT05835427
Title: The Effect of Stretching and Relaxation Exercises on Anxiety in Individuals With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Fibromyalgia
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
Keywords: exercise
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Individuals with fibromyalgia and healthy individuals will be included in the study and the effectiveness of the treatment will be examined. Within the scope of the study, relaxation and stretching exercises will be applied to both groups for eight weeks.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia individual (Experimental): Cervical Extensor Stretch, cervical flexor stretch, cervical lateral flexion stretch, thoracic stretch, pectoral stretch, lumbar extensor stretch, posterior capsule stretch, knee flexor stretch, gastro-soleus stretch, quadriceps stretch, cat-camel exercise, shoulder circles, neck flip- tilting the neck to the right and left, relaxation of the abdominal and back muscles, posterior pelvic tilt.
  Interventions: Other: Cervical Extensor Stretch
- Healthy volunteers (Experimental): Cervical Extensor Stretch, cervical flexor stretch, cervical lateral flexion stretch, thoracic stretch, pectoral stretch, lumbar extensor stretch, posterior capsule stretch, knee flexor stretch, gastro-soleus stretch, quadriceps stretch, cat-camel exercise, shoulder circles, neck flip- tilting the neck to the right and left, relaxation of the abdominal and back muscles, posterior pelvic tilt.
  Interventions: Other: Cervical Extensor Stretch

INTERVENTIONS:
Other: Cervical Extensor Stretch — Fibromyalgia individual: Within the scope of the study, relaxation and stretching exercises will be applied to both groups for eight weeks.
  Arms: Fibromyalgia individual
Other: Cervical Extensor Stretch — Healthy volunteers : Within the scope of the study, relaxation and stretching exercises will be applied to both groups for eight weeks.
  Arms: Healthy volunteers

SUMMARY:
Fibromyalgia is a non-articular, chronic rheumatic disease of unknown etiology characterized by widespread musculoskeletal pain, sleep disturbance, fatigue, and the presence of multiple tender points.

DETAILED DESCRIPTION:
Although the exact etiology cannot be determined in fibromyalgia, it is thought that there are many mechanisms that contribute to the formation of Fibromyalgia. Evidence for some biochemical, neurohormonal, central nervous system, immunological, psychological and environmental factors that may play a role in the disease has been found.

ELIGIBILITY:
Inclusion Criteria

* Volunteer
* Being diagnosed with fibromyalgia Exclusion Criteria
* Known neurological disorder
* Serious orthopedic disorders that will prevent him from exercising
* Cognitive impairment
* Using regular NSAIDs
* Being malnourished and malnourished

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 8 weeks
  In this scale filled by the patient; Physical function, feeling well, not being able to go to work, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression were measured.
  With the exception of the well-being trait, low scores indicate recovery or less affliction. Each subheading was asked to be scored between 0-10. Values of 50 points and below were considered as mildly affected, and values above 50 points were considered as severely affected.
The Pittsburg Sleep Quality Index | 8 weeks
  The Pittsburg Sleep Quality Index is a 19-item self-report scale that assesses sleep quality and impairment over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality".
Beck Anxiety Scale | 8 weeks
  It measures the frequency of anxiety symptoms experienced by the individual. It is a Likert-type self-assessment scale consisting of 21 items and scored between 0-3. The individual is asked to mark only one of the "None", "Mild", "Moderate" and "Severe" options for each item. The total score range is between 0-63. The high score total indicates the high level of anxiety experienced by the individual.
Fibromyalgia ACR Criterion assessed by Composite the Widespread Pain Scale and the Symptom Severity Scale | 8 weeks
  It is obtained by adding the Widespread Pain Scale and the Symptom Severity Scale. The maximum total score here is 19+12=31. Accordingly, scores below a total of 12 do not suggest fibromyalgia. Widespread Pain Scale ≥7 and Symptom Severity Scale ≥5.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Yoo SA, Kim CY, Kim HD, Kim SW. Effects of progressive muscle relaxation therapy with home exercise on pain, fatigue, and stress in subjects with fibromyalgia syndrome: A pilot randomized controlled trial. J Back Musculoskelet Rehabil. 2022;35(2):289-299. doi: 10.3233/BMR-191703. PMID 34151818